CLINICAL TRIAL: NCT03848598
Title: Is There a Mechanistic Reason for the Response or Non-response to Isometric Exercise in Tendinopathy?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Stijn Bogaerts, Resident staff member Physical & Rehabilitation Medicine, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: SBogaerts
Record Dates: First submitted 2019-02-13; First posted 2019-02-21 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Tendinopathy
Keywords: patellar; ultrasound; speckle; isometric
MeSH Terms: conditions — Tendinopathy; Patella Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Responders: Patients suffering from patellar tendinopathy who have complete pain resolution after performing isometric exercises.
  Interventions: Diagnostic Test: Evaluation of local tendon deformation
- Non-responders: Patients suffering from patellar tendinopathy who do not have complete pain resolution after performing isometric exercises.
  Interventions: Diagnostic Test: Evaluation of local tendon deformation

INTERVENTIONS:
Diagnostic Test: Evaluation of local tendon deformation — Ultrasound-based speckle tracking to evaluate the local tendon tissue displacement during isometric exercise.

SUMMARY:
In early phase tendinopathy, isometric exercises are seen as ideal to provide pain relief to patients. This approach is mainly based on a paper by Rio et al (2016), where they found that isometric exercises of a certain load magnitude and time (5 repetitions of 45 second hold at 70% of maximum) gave 100% pain relief for 45 minutes in patients with patellar tendinopathy. This then helps patients to perform their more heavy load exercises during rehabilitation, which would otherwise be too painful.

Unfortunately, the study of Rio et al only consisted of 6 participants, and recent papers have contradicted the findings. In Achilles tendinopathy, plantar fasciopathy and lateral elbow tendinopathy, the pain relief was not consistently present, with "responders" and "non-responders" being found in these studies. Also, a study yet to be published (poster at conference), replicating Rio et al, also found a heterogeneous response, debunking the "one size fits all" approach that seemed to work.

However, in our understanding, isometric exercises do have a crucial role in early tendinopathy management, but the way the exercise is performed, in which position, what magnitude of load, time under tension, … has an important influence. The same protocol (5 repetitions of 45 second hold at 70% of maximum) might lead to big inter-individual differences. Therefore, there might be a mechanistic reason why some patients respond, and others do not.

Fortunately, the P.I. of this current trial application has recently optimized an ultrasound-based method to quantify local tendon deformation during exercises. The main purpose of this trial is therefore to evaluate the local tendon deformation pattern of patients with tendinopathy during isometric exercises and evaluate whether there is an interindividual difference in pattern between "responders" and "non-responders".

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of patellar tendinopathy, consisting of

* pain located at the proximal part of the patellar tendon
* painful at palpation the proximal part of the patellar tendon
* Numeric Rating Scale > 1/10 with squat on decline (20°) board

Exclusion Criteria:

* previous treatment for patellar tendinopathy
* rupture of patellar tendon on ultrasound
* unclear differential diagnosis with patellofemoral pain
* concomitant neuromuscular disorders

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Patients visiting the sports medicine consultation of the University Hospitals and presenting with complaints of patellar tendinopathy will be screened for eligibility.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Local tendon tissue displacement in three layers of the tendon (deep, middle and superficial layer); as measured by ultrasound-based speckle tracking | Immediately during isometric exercise
  Millimeter

SECONDARY OUTCOMES:
Non-uniform displacement; as measured by ultrasound-based speckle tracking | Immediately during isometric exercise
  % (measure for relative displacement of the superficial layer of the tendon versus the deep layer, and then divided by the mean total displacement of the three layers combined)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No